CLINICAL TRIAL: NCT05967949
Title: A Retrospective (Non-interventional) Clinical Study on the First-line Maintenance Treatment of Peripheral T-cell Lymphoma (PTCL) With Chidamide.
Brief Title: A Retrospective Clinical Study on the First-line Maintenance Treatment of PTCL With Chidamide.
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CS123
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: PTCL
Keywords: chidamide; maintenance treatment
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: chidamide — This subset of patients received chidamide as first-line maintenance therapy.

SUMMARY:
The efficacy and safety of chidamide in first-line maintenance therapy for PTCL will be assessed through a retrospective case analysis.

DETAILED DESCRIPTION:
The study design belongs to a retrospective study, collecting information on patients with PTCL who were diagnosed and treated with chidamide as maintenance therapy at our center. The collected data includes age, gender, previous treatment regimens, results of auxiliary examinations (such as blood routine, biochemistry, bone marrow cytology, pathology, flow cytometry, NGS, etc.), as well as PET-CT images. The safety and efficacy of Chidemide as first-line maintenance therapy in PTCL will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age: 18 years and older; (2) Gender: Male/Female; (3) Diagnosed with PTCL; (4) Received chidamide as maintenance therapy after first-line treatment.

Exclusion Criteria:

* (1) Patients with other types of lymphomas; (2) Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with PTCL, who have undergone first-line treatment and are using chidemide as maintenance therapy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  progression free survival

SECONDARY OUTCOMES:
OS | 2 years
  overall survival
CR | 2 years
  complete remission
DOR | 2 years
  duration of remission

CONTACTS AND LOCATIONS:
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No